CLINICAL TRIAL: NCT06224127
Title: Treating Stress and Anxiety in Individuals With Alcohol Use Disorder (AUD) Using a Combination of TRPV-1 Channel and C-tactile Fiber Activation With Measurement of Oxytocin and Cortisol Levels
Brief Title: Treating Stress and Anxiety in Individuals With Alcohol Use Disorder (AUD)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soovu Labs Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: Soovu01-2024
Record Dates: First submitted 2024-01-15; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Anxiety Disorders; Alcohol Use Disorder; Stress, Psychological
Keywords: anxiety; Alcohol Use Disorder; stress; c-tactile fiber; heat
MeSH Terms: conditions — Anxiety Disorders; Alcoholism; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized into three groups. Group 1 receives an active heating device and placebo c-tactile fiber stimulation. Group 2 active c tactile fiber stimulation and placebo heating device. Group 3 receives active c tactile fiber stimulation and an active heating device.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subjects, assessors and investigators will not know the randomization group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Active heat and placebo c tactile stimulation (Active Comparator): Subjects will receive an active heating device and a sham c tactile stimulation device.
  Interventions: Device: active heat; Device: Sham c tactile fiber stimulation
- Placebo heat and active c tactile stimulation (Active Comparator): Subjects will receive an active c tactile stimulation device and a sham heating device.
  Interventions: Drug: Active c tactile fiber stimulation; Device: sham heat
- Active heat and active c tactile stimulation (Active Comparator): Subjects will receive an active c tactile stimulation device and an active heating device.
  Interventions: Device: active heat; Drug: Active c tactile fiber stimulation

INTERVENTIONS:
Device: active heat — Users receive an active Soovu heating pod(s).
  Arms: Active heat and active c tactile stimulation; Active heat and placebo c tactile stimulation
Drug: Active c tactile fiber stimulation — Hair brushes that activate c tactile fibers
  Arms: Active heat and active c tactile stimulation; Placebo heat and active c tactile stimulation
Device: sham heat — A Soovu heating pod(s) in the subtherapeutic temperature range
  Arms: Placebo heat and active c tactile stimulation
Device: Sham c tactile fiber stimulation — Hair brushes that do not activate c tactile fibers
  Arms: Active heat and placebo c tactile stimulation

SUMMARY:
CT fibers are found in the skin of most mammals and project to the insular cortex. Stimulation of CT fibers by light touch causes a release of oxytocin and is associated with feelings of comfort and wellbeing. Peripheral TRPV-1 channels are important in pain transmission and modulation of the stress response likely through the central release of oxytocin and are stimulated by heat. In Phase 1 investigators will test stimulation of TRPV1 channels and CT fibers in human subjects to correlate the lab findings with subjective human responses and test whether stimulation of CT fibers and TRPV-1 channels reduce anxiety and stress in subjects who suffer from AUD. Aim 1 and 2. We will define the optimal parameters for CT fiber stimulation for force, temperature, and body location. We will perform similar testing for peripheral thermal stimulation (TRPV-1) using our commercially available heating pods. Parameters tested will include the optimal body location, number of heating pods (2-4) and temperature of pods. In Aim 3 investigators will simultaneously apply both CT fiber and thermal stimulation in a proof of concept study. The experimental group will receive active CT fiber and thermal stimulation and the control group non-physiologic placebo stimulation. Subjects with a history of AUD will be randomized into control versus experimental groups and undergo stress using a validated mental calculation stressors. Stress, cravings, and anxiety will be measured using standardized assessments, and investigators will measure salivary oxytocin and cortisol levels, potentially biomarkers.

DETAILED DESCRIPTION:
36 subjects with a history of AUD within the past six months will be recruited for this study. Subjects will be randomized into three groups. Group 1 receives an active heating device and placebo c-tactile fiber stimulation. Group 2 active c tactile fiber stimulation and placebo heating device. Group 3 receives active c tactile fiber stimulation and an active heating device. All subjects will have baseline labs drawn, then undergo 10 minutes of experimental stimulation according to group number 1,2 or 3,After 10 minutes, subjects will be given a validated experimental stressor that takes approximately 15 minutes. During this time, subjects will also receive the experimental stimulation per their experimental group After the experimental stress is concluded, stimulation will continue for an additional 5 minutes. Oxytocin and cortisol via salivary samples will be collected throughout and at the conclusion of the trial. Subjects will be followed for one hour post trial. Both laboratory testing and assessment measures will be repeated at 30 and 60 minutes post experimental treatment. Assessment measures include the VAS-A, the PROMIS anxiety short form, and the desires for alcohol questionnaire. The active placebo is thermal stimulation at 37°C over the trapezius using the same number of heating pods. Placebo CT stimulation will occur by placing the von Frey filaments, which provide two standard deviations less than the optimal pressure. Subjects will not be informed about which group they were randomized into.

ELIGIBILITY:
Inclusion Criteria:

* A history of AUD within the past six months

Exclusion Criteria:

Unstable medical or psychological status

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety rating | at baseline and every 15 minutes during the study and for 90 minutes post study
  Patient-Reported Outcomes Measurement Information System anxiety short form, 0-10 with 10 meaning more anxiety and 0 no anxiety
anxiety level | at baseline and every 15 minutes during the study and for 90 minutes post study
  Visual analogue scale for anxiety. 0-10 with 10 meaning more anxiety and 0 no anxiety
desires for alcohol questionnaire | at baseline and every 30 minutes during the study and for 90 minutes post study
  desires for alcohol questionnaire

SECONDARY OUTCOMES:
Oxytocin | Baseline and every 15 minutes during the study and for 90 minutes post study
  oxytocin levels
cortisol levels | Baseline and every 15 minutes during the study and for 90 minutes post study
  salivary cortisol

CONTACTS AND LOCATIONS:
Overall Officials: charles chabal, MD, Principal Investigator — soovu labs
Locations (1):
- Soovu Labs Inbc., Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data records will be available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: At study conclusion and for 5 years

REFERENCES:
- See also: description of heating device — http://soovu.com